CLINICAL TRIAL: NCT04471285
Title: Acupuncture as a Treatment for Symphysiolysis Pain and Ability in Pregnant Women.
Brief Title: Symphysiolysis: Acupuncture Therapeutic Benefits: a Randomized Placebo Controlled Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, jaffea, OBGYN resident, MD MPH, Shaare Zedek Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0115-18-SZMC
Record Dates: First submitted 2020-07-02; First posted 2020-07-15 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Single Embryo Pregnancy; Gestational Weeks 24-42; Pain/Sensitivity >5 on Numeric Rating Scale (NRS)
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The trial doctor will mark the woman's chart with a continuous number that will become her number in the trial, and she will then be referred to the acupuncturist. , she will receive an acupuncture treatment according to the randomized numbers for acupuncture V or acupuncture P. Approximately 30 minutes after the acupuncture treatment began, the woman will be asked once again to assess her level of pain. An improvement of 1.5 marks on the NRS scale is considered a positive response. Women whose response after 30 minutes of acupuncture is less than this will be given the opposite acupuncture treatment. Those who received V acupuncture will receive P acupuncture and those who received P acupuncture will receive V acupuncture. A woman will be called again if her pain is significantly worse. She will then receive the treatment that has been found most effective between the two acupuncture treatments she received previously.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- true acupuncture (Active Comparator): patient will get treatment according to the point the will help the symphysiolysis according to the Alternative medicine
  Interventions: Procedure: acupuncture
- Sham acupuncture (Sham Comparator): patient will get treatment according to the point the will NOT help the symphysiolysis according to the Alternative medicine
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: acupuncture — acupuncture
  Arms: true acupuncture
Procedure: Sham acupuncture — Sham acupuncture
  Arms: Sham acupuncture

SUMMARY:
a randomized, observer blind and placebo-controlled cross-over study in which true acupuncture (Verum)(V) was compared to "placebo" acupuncture (P).

the investigators evaluate the effect of the acupuncture on the pain and the ability of the pregnant patient.

DETAILED DESCRIPTION:
the investigators recruit women who diagnose with symphysiolisis by having 2 out of 3 of the follow:

* Examine for pain or sensitivity to touch on pubic symphysis joint.
* Modified Trendelenburg's test
* Active straight leg raise test The trial doctor will mark the woman's chart with a continuous number that will become her number in the trial, and she will then be referred to the acupuncturist.

Women will be randomly divided at a 1:1 ratio, according to the randomized number chart prepared by the trial's statistician. The list of random numbers will be delivered to the head of the acupuncturist team and it will be the only copy in existence aside from the one belonging to the statistician. According to that list of numbers, the head acupuncturist will instruct the acupuncturist on call as to the type of acupuncture to be performed, true (V) vs. placebo (P) on the participant . The type of acupuncture (V or P) will be recorded in the woman's chart.

The treatment will be conducted by one of the acupuncturists on staff at the integrative medical center. All the acupuncturists have many years of experience in treating pregnant women with Chinese medicine. The acupuncture will be carried out with 0.18/40mm single use needles. Point selection and numbers of points used will be determined following the evaluation of the acupuncturist according to the accepted standards of in Chinese medicine. They will not, however, deviate from the list of true acupuncture points in the list of possible true paints . Placebo acupuncture will be three to four points selected at random from the list of placebo points . The acupuncturist's evaluation in the placebo group will be the same as in the evaluation in the treatment group and the true acupuncture points selected during that time will be the ones used in case of failure and continued pain following the first (placebo) treatment, after cross over.

It should be noted that the woman's assessment and the exam will take place before the acupuncture treatment begins, whether it is the true or placebo group.

Approximately 30 minutes after the acupuncture treatment began, the woman will be asked once again to assess her level of pain. An improvement of 1.5 marks on the NRS scale is considered a positive response. Women whose response after 30 minutes of acupuncture is less than this will be given the opposite acupuncture treatment. Those who received V acupuncture will receive P acupuncture and those who received P acupuncture will receive V acupuncture. A woman will be called our team if her pain is significantly worse. She will then receive the treatment that has been found most effective between the two acupuncture treatments she received previously.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years
* Single embryo pregnancy in week 24-42
* was diagnosed with symphysiolisis according to written above
* Pain/sensitivity >5 on NRS scale in symphysis pubis area for more than two weeks

Exclusion Criteria:

* Lack of proficiency in Hebrew or English
* Pain from a different source
* pelvic bone disease or history of severe pelvic bone injury
* Thrombocytopenia (plt<50.000)
* Acupuncture treatment is contraindicated
* High risk pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
pain improvement | 30 minutes
  improvement of 1.5 marks on the Numeric Rating Scale (NRS) ( 0-10 , 0=no pain, 10=worst pain) as describe by the patient.

SECONDARY OUTCOMES:
improvement in the ability by using Modified Oswestry Disability Questionnaire (MODQ) - Questionnaire | 48-72 hours
  To compare the functional effects of true and Sham acupuncture on the daily activities/ ability of women with symphysiolysis. the Questionnaire check the daily function of 10 daily activity's ( Pain Intensity ,Personal Care (e.g., Washing, Dressing) Lifting,Walking,Sitting,Standing,Sleeping,Social Life,Traveling,Employment / Homemaking).
  For each section the total possible score is 5: if the first statement - witch represent no restriction -is marked the section score = 0, if the last statement is marked-witch represen severe disability the score is 5.
  the total score number is calculated by : Score: /50 x 100 = ____% points Example: 16 (total scored-by the patient answers)/ 50 (total possible score) x 100 = 32%

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, MD, Principal Investigator — head of alternative medicine; Sorina Grisaro, MD PhD, Study Director — head of OBGYN department
Locations (1):
- Shari Zedek Medical Center, Jerusalem, Israel